CLINICAL TRIAL: NCT00784160
Title: Study for Dermatological Evaluation of Topic Compatibility (Primary and Accumulated Dermical Irritability, Dermical Sensitivity) of Dermacyd PH_DETINBACK Tangerine Mix.
Brief Title: Dermacyd PH_DETINBACK Tangerine Mix (Lactic Acid)- Compatibility
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: LACAC_L_04308
Record Dates: First submitted 2008-10-31; First posted 2008-11-03 (Estimated); Last update posted 2009-08-25 (Estimated); Status verified 2009-08

CONDITIONS: Hygiene
MeSH Terms: interventions — Lactic Acid

ARMS (1):
- 1 (Experimental): Lactic Acid
  Interventions: Drug: Lactic Acid (Dermacyd PH_DETINBACK Tangerine Mix)

INTERVENTIONS:
Drug: Lactic Acid (Dermacyd PH_DETINBACK Tangerine Mix) — Lactic Acid

SUMMARY:
The purpose of this study is to demonstrate the absence of irritation potential (primary dermic irritability and cumulated dermic irritability) and allergy (sensibilization) of the product Dermacyd PHDETINBACK Tangerine Mix (Lactic Acid).

ELIGIBILITY:
Inclusion criteria:

* Age between 18 and 60 years old;
* Phototype Skin I,II, III e IV;
* Integral skin test in the region;
* Willingness in following the study procedures and to be present in the clinic at the days and scheduled time for medical evaluations and for application of occlusion;

Exclusion criteria:

* Lactation or gestation;
* Personnel history of atopy;
* History of sensitivity or irritation for topic products;
* Active cutaneous disease;
* Use of new drugs or cosmetics during the study;

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2008-07; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
The absence of primary and accumulated dermical irritability and dermical sensitivity will be evaluated using International Contact Dermatitis Research Group (ICDRG) scale. | Throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Jaderson Lima, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, São Paulo, Brazil